CLINICAL TRIAL: NCT03665831
Title: Treatment of Comorbid Depression and Cognitive Impairment in Older Adults With Neurocognitive Disorders Using Deep Transcranial Magnetic Stimulation (dTMS)
Brief Title: Deep TMS for Comorbid Depression and Cognitive Impairment in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Brainsway (Industry); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Linda Mah, MD, Clinician Scientist, Rotman Research Institute at Baycrest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICP-2-00095
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder; Alzheimer Disease; Mild Cognitive Impairment
Keywords: dTMS; depression; magnetic; iTBS
MeSH Terms: conditions — Depressive Disorder, Major; Alzheimer Disease; Cognitive Dysfunction; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Active H1 Coil deep rTMS active treatment (Experimental)
  Interventions: Device: Brainsway H1-Coil Deep TMS System

INTERVENTIONS:
Device: Brainsway H1-Coil Deep TMS System — Deep Transcranial Magnetic Stimulation (dTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel dTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions. dTMS will be administered daily for 4 consecutive weeks.

SUMMARY:
In this study, the investigators will be examining the effects of the deep repetitive transcranial magnetic stimulation (rTMS) using the H1 coil in patients over the age of 60 diagnosed with mild to early-moderate Alzheimer's disease (AD) or mild cognitive impairment (MCI) and comorbid Major Depressive Disorder (MDD) who have been unable to tolerate or failed to respond to antidepressant medications. The coil was designed to stimulate deeper regions of the left dorsolateral prefrontal cortex (DLPFC). Based on prior research, the investigators propose that active stimulation with the H1 coil for 4 weeks may result in significant remission rates and will be tolerable and safe.

DETAILED DESCRIPTION:
This study is an open-label trial to evaluate the safety and efficacy of H1-coil dTMS in treating depression in MCI and mild AD patients over 60 years of age who have not tolerated or failed to respond to antidepressant medications. 28 patients will be assigned to receive 4 consecutive weeks of daily active dTMS treatment. The long-term effects of treatment on emotional cognitive measures will be assessed at a 4-week follow-up visit (8 weeks from baseline). Symptom change and remission criteria will be assessed using the Montogmery-Asberg Depression Rating Scale (MADRS). Cognition will be assessed using a validated neuropsychological battery.

We will also offer patients to receive 4 weeks of treatment using theta-burst TMS, which is a milder version of TMS.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM 5 criteria for Major or Mild Neurocognitive Disorder due to Alzheimer's disease with Clinical Dementia Rating Scale (CDR) score of at least 0.5
* have been diagnosed with DSM5 Major Depressive Disorder, with the current episode longer than 4 weeks but less than 5 years
* did not respond to or did not tolerate antidepressant treatment
* are willing to provide informed consent
* are able to follow the treatment schedule
* are stable on medications for 2 months and are not expected to change medication during the entire study period (if they are taking medications)
* have a satisfactory safety screening questionnaire for TMS
* have an informant/study partner who is able to complete study questionnaires regarding the participant

Exclusion Criteria:

* have a metal plate in their head, except in the mouth (such as an ear implant, implanted brain stimulators, aneurysm clips)
* have known increased pressure or a history of increased pressure in their brain, which may increase their risk for having seizures
* have a cardiac pacemaker
* have an implanted medication pump
* have a central venous line
* have a significant heart disease or history of stroke
* Modified Hachinski Score (MHIS) > 3 (to exclude those with significant vascular component to memory loss)
* have a history of any psychotic disorder, bipolar disorder, eating disorder, obsessive compulsive disorder, post-traumatic stress disorder, or dementia other than AD
* have a history of substance abuse in the last 6 months
* have a history of stroke or other brain lesions
* have a personal history of epilepsy
* have a family history of epilepsy
* are a pregnant or breast-feeding woman
* are taking psychotropic medications including antidepressant medications, antipsychotics or mood stabilizing medications due to increased risk of seizure
* are taking memantine
* have a history of abnormal MRI of the brain
* have significant hearing loss requiring use of hearing aids
* have untreated hypo- or hyper-thyroidism

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) | 4 weeks
  Therapeutic efficacy will be evaluated with the MADRS, a 10-item checklist. An effect size (Cohen's d) of 0.5 will be considered a minimally important effect size.

SECONDARY OUTCOMES:
Remission Rates Compared Within Treatment Group | 4 weeks
  Remission defined as MADRS < 10.
Response Rates Compared Within Treatment Group | 4 weeks
  Response rate refers to the percentage of patients who responded to dTMS treatment and response is defined as a ≥50% reduction in MADRS score from baseline.
Change From Baseline on the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | 4 weeks
  This 16-item questionnaire is designed to help assess the degree of enjoyment and satisfaction experienced during the past week. Administration time is approximately 5 minutes.
Change From Baseline on the Neuropsychological Battery | 4 weeks
  Cognitive scores from the neuropsychological battery at baseline will be compared to 4 weeks post-intervention Cognitive domains tested include executive function, memory, language, attention, and intelligence.
Change in Functional Connectivity between PFC and Limbic Regions | 4 weeks
  Subjects will have magnetic resonance imaging (MRI) scans of the brain. The change in functional connectivity between PFC and limbic regions, and within the default mode network, at rest is measured using resting state fMRI.
Change in Perfusion within Prefrontal Cortex (PFC) and Posterior Cingulate Cortex (PCC) | 4 weeks
  Measured using Arterial Spin Labeling (ASL) fMRI scan.
Change in frontal theta power within the Anterior Cingulate Cortex (ACC) | 4 weeks
  Measured with electroencephalography (EEG) and/or magnetoencephalography (MEG).

CONTACTS AND LOCATIONS:
Locations (1):
- Rotman Research Institute at Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hodzic-Santor BH, Meltzer JA, Verhoeff NPLG, Blumberger DM, Mah L. Safety, tolerability, and feasibility of deep transcranial magnetic stimulation for late-life depression with comorbid major or mild neurocognitive disorder. Int Psychogeriatr. 2021 Jan;33(1):99-101. doi: 10.1017/S1041610220003543. Epub 2020 Nov 6. No abstract available. PMID 33153503